CLINICAL TRIAL: NCT02531945
Title: Scoliosis Patients Aged 10-13 Years: Monitoring of Scoliosis by the Surface Topography
Brief Title: Evaluation of the Surface Topography for Monitoring Scoliosis Patients Aged 10-13 Years
Acronym: SCOBIOMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/14/7419
Record Dates: First submitted 2015-08-18; First posted 2015-08-25 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2018-05

CONDITIONS: Scoliosis
Keywords: topography; cobb angle
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): The device used in this research to the topography examination is three-dimensional morphometry device of AXS Medical society : the BIOMOD L.
  'Use of Biomod device' for all the patient in addition to the conventional X-ray examination.
  Interventions: Device: Use of Biomod device

INTERVENTIONS:
Device: Use of Biomod device

SUMMARY:
The main objective of the study is to investigate the correlation between the measurement of the Cobb angle (angle of scoliosis) by conventional radiography and angle measured by surface topography.

The device used in this research to the topography examination is three-dimensional morphometry device of AXS Medical society : the BIOMOD L.

DETAILED DESCRIPTION:
For usual follow-up visit, patients will have a x-ray examination of the spine and the surface topography. The measurement of the angle of scoliosis is achieved by two independent operators for both methods.

Patients then have a follow-up visit at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with idiopathic scoliosis,
* Body mass index BMI below or equal to 25,
* Cobb angle measured on radiographs between 10 and 25 degrees,
* Parental authorization.

Exclusion Criteria:

* Patient with secondary scoliosis (neurological, Prader Willi syndrome...)

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation between the measurement of Cobb angle by conventional .radiography and surface topography. | up to 1 year
  Number of participants with the same cobb angle measured by surface topography and measured by x-ray.

SECONDARY OUTCOMES:
Reproducibility within the operator of measurement of the angle by surface topography | At each visit two successive measurements are made by the operator for the same patient. up to 1 year
  up to 1 year
Reproducibility between the operator of measurement of the angle by surface topography | up to 1 year
  Two independent operators will measures.
The sensitivity of the topography on the detection of the deterioration of the Cobb angle | up to 1 year
  The sensitivity of the surface topography to detect a worsening of one year more than 5 ° C over the Cobb angle will be assessed compared to the radiograph. It will be obtained by the ratio between the number of aggravations detected by the surface topography and the total number of exacerbations diagnosed by radiography.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme SALES DE GAUZY, Principal Investigator — UH Toulouse
Locations (1):
- UH toulouse, Toulouse, France

REFERENCES:
- [Result] Bolzinger M, Bernardini I, Thevenin Lemoine C, Gallini A, Accadbled F, Sales de Gauzy J. Monitoring adolescent idiopathic scoliosis by measuring ribs prominence using surface topography device. Spine Deform. 2021 Sep;9(5):1349-1354. doi: 10.1007/s43390-021-00327-1. Epub 2021 Mar 29. PMID 33782905